CLINICAL TRIAL: NCT06599840
Title: Improving Self-management in Childhood Diabetes - Feasibility and Preliminary Effects of a CBT-based Intervention for Parents
Brief Title: Feasibility Study of a Behavioral Parent Intervention to Support Self-management in Pediatric Typ 1 Diabetes
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Collaborators: Karolinska University Hospital (Other)
Responsible Party: Principal Investigator, Brjann Ljotsson, Professor, licensed psychologist, Karolinska Institutet
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Dnr2021-01558_feasibility
Record Dates: First submitted 2024-09-09; First posted 2024-09-19 (Actual); Last update posted 2025-08-27 (Actual); Status verified 2025-08

CONDITIONS: Type 1 Diabetes Mellitus; Parent-Child Relations; Self-management; Behavioral Intervention
Keywords: feasibility study; type 1 diabetes; diabetes self-management; parent support; parent intervention; pediatric self-management; behavioral intervention; pediatric type 1 diabetes; self-management problems; parent training; CBT; T1D; self-management intervention
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention group (Other): CBT-based parent intervention consisting of 7 group sessions.
  Interventions: Behavioral: Parent intervention

INTERVENTIONS:
Behavioral: Parent intervention — This is a novel intervention based on established CBT-based parenting strategies that are regularly used to strengthen parent-child cooperation and reduce conflicts. Here, the strategies are adapted to address typical challenges of T1D family life. The program structure consists of six weekly modules and a seventh booster module. Each of the first six modules has a theme with information on a parental strategy associated with the theme, self-reflective questions, and an assignment where parents plan to implement the strategy during the upcoming week. One month later, a seventh session is held to summarize the program and make plans for future progress.

SUMMARY:
This study investigates feasibility and preliminary effects of a new behavioral parent intervention that aims to support and improve pediatric diabetes self-management

DETAILED DESCRIPTION:
Diabetes self-management is extensive, complex and places high demands on the affected individual and his/her family. Today, half of Swedish children and adolescents with type 1 diabetes (T1D) do not reach target levels of glycemic control. Among the various factors that influence glycemic control, family function is of great importance. Parent-child conflicts surrounding self-management tasks have been shown to predict glycemic control deterioration over time. This study will explore feasibility and preliminary effects of a new behavioral parent intervention that aims to strengthen parent-child cooperation and facilitate diabetes routines in every-day-life. The results of the feasibility study will guide further refinement of the intervention, and the design of a future RCT.

Through digital ads and posters at the diabetes clinics in Stockholm, we will recruit parents of children aged 9-14 with T1D experiencing problems in getting diabetes self-management routines to work in every-day-life. The intervention is held at the hospital and includes six weekly group sessions and a booster session one month later. At the end of each session, parents plan to use a new behavioral strategy at home during the upcoming week. This feasibility study will explore participant satisfaction and attendance combined with qualitative assessments of their experiences. Preliminary effects are investigated through repeated assessments of a set of digitalized questionnaires, data from the national diabetes registry and online blood glucose data during the intervention phase, post intervention and at 3- months follow up.

This intervention is believed to be an effective way to target and prevent T1D self-management problems and may come to serve as an important complement to standard diabetes treatment.

ELIGIBILITY:
Inclusion Criteria:

* Parents/guardians of children aged 9-14 with type 1 diabetes.
* The child has had type 1 diabetes for at least one year.
* The parent experience difficulties in managing daily life and/or the parent-child collaboration around self-management routines.
* The perceived difficulties should not solely be due to perceived problems in the medical aspects of the diabetes treatment, such as a perceived need for more support in insulin dosing, more diabetes education, or technical/medical support. This criterion is based solely on the subjective judgement of the parent him-/herself.
* The child receives diabetes care at one of the three diabetes clinics in the Stockholm Region.
* The parent speaks, understands, and can read Swedish.
* The parent claims to be motivated and has the practical possibility to participate in the study and attend group meetings.

Exclusion Criteria:

* The parent reports current and severe psychiatric conditions in themselves or the child that need to be prioritized, such as severe depression, suicidal thoughts/self-harm, psychosis, or mania.
* The parent is involved in another psychological treatment of a behavior-changing nature that is in an active phase, either concerning themselves or a child.
* Major planned changes in diabetes treatment that require learning and behavioral changes, such as transitioning from pen to pump, and that are expected to occur during the first 3.5 months of the study (active intervention phase).

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2024-09-20 (Actual); Primary Completion 2025-08-19 (Actual); Study Completion 2025-11-01 (Estimated)

PRIMARY OUTCOMES:
Diabetes Treatment Satisfaction Questionnaire - parent report | From baseline until 26 weeks.
  This is a 14 item questionnaire that aim to measure parental satisfaction with the diabetes treatment. Parents are asked to rate their satisfaction on a likert scale from 0 = very unsatisfied, to 6 = very satisfied about a range of diabetes treatment domains. The questionnaire is based on the adult version of DTSQ and adapted to pediatric type 1 diabetes. Translated to Swedish and validated in a Swedish cohort.
Diabetes Treatment Satisfaction Questionnaire - parent report | From baseline until 15 weeks.
  This is a 14 item questionnaire that aim to measure parental satisfaction with the diabetes treatment. Parents are asked to rate their satisfaction on a likert scale from 0 = very unsatisfied, to 6 = very satisfied about a range of diabetes treatment domains. The questionnaire is based on the adult version of DTSQ and adapted to pediatric type 1 diabetes. Translated to Swedish and validated in a Swedish cohort.
Diabetes Treatment Satisfaction Questionnaire - parent report | Weekly from baseline to 14 weeks
  This is a 14 item questionnaire that aim to measure parental satisfaction with the diabetes treatment. Parents are asked to rate their satisfaction on a likert scale from 0 = very unsatisfied, to 6 = very satisfied about a range of diabetes treatment domains. The questionnaire is based on the adult version of DTSQ and adapted to pediatric type 1 diabetes. Translated to Swedish and validated in a Swedish cohort.

SECONDARY OUTCOMES:
Glycaemic control | From baseline until 26 weeks.
  HbA1c values taken during diabetes clinic visits, registered in the national diabetes registry.
DISABKIDS (child QoL) - parent report | From baseline until 26 weeks.
  This is a questionnaire that aims to measure health related quality of life in children living with chronic conditions. The parent version comprises 37 items concerning aspects of how the condition may affect the child in every-day-life, such as whether the child is worried about his/her future, if he/she spends time with friends. It is scored using five ordinal response categories ranging from "never" to "always." The negative oriented items are coded 4 ("never") to 0 ("always") whereas the positive oriented questions are inverted, so that higher score indicates higher quality of life.
Days of physical activity | From baseline until 26 weeks.
  Number of day per week of physical activity. Information taken during diabetes clinic visits, and registered in the national diabetes registry.
PedsQL - Family Impact Measure (parent QoL) | From baseline until 26 weeks.
  This instrument measures quality of life for parents who have children with a chronic disorder. It includes 36 items concerning physical, emotional, social and cognitive functions as well as daily activities, family relations, communication and family worry. Items are answered on a five-grade scale from 0 = never a problem, to 4 = almost always a problem. These result for each item is transformed so that 0 = 100, 1 = 75, 2 = 50, 3 = 25, 4 = 0, and the sum score is divided by the number of items, so that higher score indicates higher quality of life.
Me As Parent | From baseline until 26 weeks.
  This is a 16-item measure that aim to measure aspects of parenting self-regulation, representing the degree to which participants perceive themselves as efficacious and competent in their role as parents. The scale includes 16 items covering the four subdomains of self-efficacy, personal agency, self-sufficiency and self-management. Items are rated on a scale from 1 = strongly disagree, to 5 = strongly agree.
Getting Self-Management Routines Done | From baseline until 26 weeks.
  This 2-item questionnaire is developed by the research group and aims to serve as a parent-reported proxy for the two key self-management behaviors: taking insulin and handling high and low blood glucose values. In percentages from 0-100%, parents are asked to estimate to what extent their child 1) takes insulin and 2) handles high and low blood glucose values, in relation to all the times these behaviors are required.
Parental Challenges in Diabetes Self-Management | From baseline until 26 weeks.
  This questionnaire is developed by this research group and based on common diabetes-specific themes of parental, behavioral challenges reported by parents in an interview study conducted by the group. In 12 items, parents are asked to rate how often they experience a set of challenges on a Likert scale from 0 = never, to 4 = always. These items cover four domains 1) parent worry and frustration, 2) talking, asking and reminding 3) child resistance to self-management routines, 4) child resistance to communication about self-management. This is a pilot use of the questionnaire, testing the items before deciding on future validation and psychometric evaluation. We will also use it to look at participants responses over time at a qualitative, clinical and explorative level and to investigate how the domains relate to eachother, to glycemic control and how/if responses change over time.
General Anxiety Disorder -7 | From baseline until 26 weeks.
  This 7-item version of the GAD questionnaire is a short measure of symptoms of anxiety. Participants are asked how often they have been bothered by a set of anxiety symptoms the last 2 weeks ranging from 0=not at all, to 7=daily. The measure will serve as a control variable in mediation analyses.
Diabetes Family Conflict Scale - parent | From baseline until 26 weeks.
  This 15-item questionnaire targets family conflicts about diabetes self-management tasks. Parents are asked how often they argue with their children about a range of different self-management routines on a scale from 0=never, 1=sometimes and 2=almost always. The sum score is multiplied by 50 giving a maximum score of 100. The last update of the English version from 2023 was translated into Swedish by this research team in 2024.
Perceived Stress Scale 10 | From baseline until 26 weeks.
  This is the 10 item version of the standardized measurement of stress, the PSS-10. Participants are asked how often they have experienced a set of stress symptoms during the last month, ranging from 0=never to 4=very often.
Parenting Practices Scale | From baseline until 26 weeks.
  Parents answer six questions about parenting practices over the last two weeks. Items are rated on a seven point Likert scale from 'Never' (coded as 1) to 'Many times a day' (coded 7), resulting in a range of 6-42 with higher scores indicating greater use of parenting skills.
Time in Target (TiT) | From baseline until 26 weeks.
  TiT is the percentage of time that blood glucose levels have been within the target interval 4-8 mmol/l during the last 2 weeks.
  This data will be taken from the national diabetes registry (NDR), and via the Glooko online glucose system.
Mean glucose level | From baseline until 26 weeks.
  The mean glucose level during the past 2 weeks. This data will be taken from the national diabetes registry (NDR), and gathered via the Glooko online glucose system.
Blood glucose variation | From baseline until 26 weeks.
  Standard deviation of blood glucose levels during the past 2 weeks. This data will be taken from the national diabetes registry (NDR), and gathered via the Glooko online glucose system.
Time with low blood glucose | From baseline until 26 weeks.
  Percentage of time during the past two weeks when blood glucose values have reached below 3 mmol/l. This data will be gathered via the Glooko online glucose system.
Ketoacidosis | From baseline until 26 weeks.
  Number of incidents of ketoacidosis as registered in the national diabetes registry.
Severe hypoglycemia | From baseline until 26 weeks.
  Number of incidents of hypoglycemia as registered in National Diabetes Registry.
Visits at the diabetes clinic | From baseline until 26 weeks.
  Number of visits registered at the National Diabetes Registry.
Client Satisfaction Questionnaire - 8 | 15 weeks after baseline
  CSQ is a cross-treatment questionnaire that aims to measure patient-reported satisfaction with the treatment they have received. This version of the CSQ includes 8 items that ask participants to rate their satisfaction on a 4-point scale where higher scores indicates higher satisfaction.
DISABKIDS (child QoL) generic + diabetes module - child report | From baseline until 15 weeks.
  This is a 37 item questionnaire that aims to measure health related quality of life in children living with chronic conditions. Added to this questionnaire is the diabetes module with 10 diabetes-specific items. Questions concern aspects of how often the condition affects different aspects of every-day-life, such as whether the child feels lonely due to his/her condition, or if he/she is bothered by the medical treatment. It is scored using five ordinal response categories ranging from "never" to "always." The negative oriented items are coded 4 ("never") to 0 ("always") whereas the positive oriented questions are inverted, so that higher score indicates higher health related quality of life.
Diabetes Family Conflict Scale - youth report | From baseline until 15 weeks.
  This 15-item questionnaire targets family conflicts about diabetes self-management tasks. Children/adolescents are asked how often they argue with their parents about a range of different self-management routines on a scale from 0=never, 1=sometimes and 2=almost always. The sum score is multiplied by 50 giving a maximum score of 100, with a higher score indicating more conflicts. The last update of the English version from 2023 was translated into Swedish by this research team in 2024.
Time with high blood glucose | From baseline until 15 weeks.
  Percentage of time the past 2 weeks when blood glucose levels have reached above 13.9 mmol/l. This data will be gathered via the Glooko online glucose system.
Glycaemic control | From baseline until 15 weeks.
  HbA1c values taken during diabetes clinic visits, registered in the national diabetes registry.
Days of physical activity | From baseline until 15 weeks.
  Number of day per week of physical activity. Information taken during diabetes clinic visits, and registered in the national diabetes registry.
DISABKIDS (child QoL) - parent report | From baseline until 15 weeks.
  This is a questionnaire that aims to measure health related quality of life in children living with chronic conditions. The parent version comprises 37 items concerning aspects of how the condition may affect the child in every-day-life, such as whether the child is worried about his/her future, if he/she spends time with friends. It is scored using five ordinal response categories ranging from "never" to "always." The negative oriented items are coded 4 ("never") to 0 ("always") whereas the positive oriented questions are inverted, so that higher score indicates higher quality of life.
PedsQL - Family Impact Measure (parent QoL) | From baseline until 15 weeks.
  This instrument measures quality of life for parents who have children with a chronic disorder. It includes 36 items concerning physical, emotional, social and cognitive functions as well as daily activities, family relations, communication and family worry. Items are answered on a five-grade scale from 0 = never a problem, to 4 = almost always a problem. These result for each item is transformed so that 0 = 100, 1 = 75, 2 = 50, 3 = 25, 4 = 0, and the sum score is divided by the number of items, so that higher score indicates higher quality of life.
Me As Parent | From baseline until 15 weeks.
  This is a 16-item measure that aim to measure aspects of parenting self-regulation, representing the degree to which participants perceive themselves as efficacious and competent in their role as parents. The scale includes 16 items covering the four subdomains of self-efficacy, personal agency, self-sufficiency and self-management. Items are rated on a scale from 1 = strongly disagree, to 5 = strongly agree.
Getting Self-Management Routines Done | From baseline until 15 weeks.
  This 2-item questionnaire is developed by the research group and aims to serve as a parent-reported proxy for the two key self-management behaviors: taking insulin and handling high and low blood glucose values. In percentages from 0-100%, parents are asked to estimate to what extent their child 1) takes insulin and 2) handles high and low blood glucose values, in relation to all the times these behaviors are required.
Parental Challenges in Diabetes Self-Management | From baseline until 15 weeks.
  This questionnaire is developed by this research group and based on common diabetes-specific themes of parental, behavioral challenges reported by parents in an interview study conducted by the group. In 12 items, parents are asked to rate how often they experience a set of challenges on a Likert scale from 0 = never, to 4 = always. These items cover four domains 1) parent worry and frustration, 2) talking, asking and reminding 3) child resistance to self-management routines, 4) child resistance to communication about self-management. This is a pilot use of the questionnaire, testing the items before deciding on future validation and psychometric evaluation. We will also use it to look at participants responses over time at a qualitative, clinical and explorative level and to investigate how the domains relate to eachother, to glycemic control and how/if responses change over time.
General Anxiety Disorder -7 | From baseline until 15 weeks.
  This 7-item version of the GAD questionnaire is a short measure of symptoms of anxiety. Participants are asked how often they have been bothered by a set of anxiety symptoms the last 2 weeks ranging from 0=not at all, to 7=daily. The measure will serve as a control variable in mediation analyses.
Diabetes Family Conflict Scale - parent | From baseline until 15 weeks.
  This 15-item questionnaire targets family conflicts about diabetes self-management tasks. Parents are asked how often they argue with their children about a range of different self-management routines on a scale from 0=never, 1=sometimes and 2=almost always. The sum score is multiplied by 50 giving a maximum score of 100. The last update of the English version from 2023 was translated into Swedish by this research team in 2024.
Perceived Stress Scale 10 | From baseline until 15 weeks.
  This is the 10 item version of the standardized measurement of stress, the PSS-10. Participants are asked how often they have experienced a set of stress symptoms during the last month, ranging from 0=never to 4=very often.
Time in Target (TiT) | From baseline until 15 weeks.
  TiT is the percentage of time that blood glucose levels have been within the target interval 4-8 mmol/l during the last 2 weeks.
  This data will be taken from the national diabetes registry (NDR), and will also be gathered repeatedly during the intervention via the Glooko online glucose system.
Visits at the diabetes clinic | From baseline until 15 weeks.
  Number of visits registered at the National Diabetes Registry.
Parenting Practices Scale | From baseline until 15 weeks.
  Parents answer six questions about parenting practices over the last two weeks. Items are rated on a seven point Likert scale from 'Never' (coded as 1) to 'Many times a day' (coded 7), resulting in a range of 6-42 with higher scores indicating greater use of parenting skills.
Parental Challenges in Diabetes Self-Management | Weekly from baseline to 14 weeks.
  This questionnaire is developed by this research group and based on common diabetes-specific themes of parental, behavioral challenges reported by parents in an interview study conducted by the group. In 12 items, parents are asked to rate how often they experience a set of challenges on a Likert scale from 0 = never, to 4 = always. These items cover four domains 1) parent worry and frustration, 2) talking, asking and reminding 3) child resistance to self-management routines, 4) child resistance to communication about self-management. This is a pilot use of the questionnaire, testing the items before deciding on future validation and psychometric evaluation. We will also use it to look at participants responses over time at a qualitative, clinical and explorative level and to investigate how the domains relate to eachother, to glycemic control and how/if responses change over time.
Getting Self-Management Routines Done | Weekly from baseline to 14 weeks
  This 2-item questionnaire is developed by the research group and aims to serve as a parent-reported proxy for the two key self-management behaviors: taking insulin and handling high and low blood glucose values. In percentages from 0-100%, parents are asked to estimate to what extent their child 1) takes insulin and 2) handles high and low blood glucose values, in relation to all the times these behaviors are required.
Mean glucose level | From baseline until 15 weeks.
  The mean glucose level during the past 2 weeks. This data will be taken from the national diabetes registry (NDR), and gathered via the Glooko online glucose system.
Blood glucose variation | From baseline until 15 weeks.
  Standard deviation of blood glucose levels during the past 2 weeks. This data will be taken from the national diabetes registry (NDR), and via the Glooko online glucose system.
Time with low blood glucose | From baseline until 15 weeks.
  Percentage of time during the past two weeks when blood glucose values have reached below 3 mmol/l. This data will be gathered via the Glooko online glucose system.
Ketoacidosis | From baseline until 15 weeks.
  Number of incidents of ketoacidosis registered in the National Diabetes Registry.
Severe hypoglycemia | From baseline until 15 weeks.
  Number of incidents of hypoglycemia as registered in National Diabetes Registry.
Short Engagement Questionnaire | Weekly from baseline until 14 weeks.
  This questionnaire is newly developed by the research group and is to be piloted in the current study. The length of questionnaire is adapted to individual CBT treatments depending on the number of treatment components that are presented. One week after a new behavioral strategy and an associated assignment have been presented to the participants, they are asked to rate their engagement according to the following three domains:
  1. Frequency: how many days they have used the strategy (1 - 7),
  2. Intensity: how much effort they have put down in using it (0 = none, to 5 = a lot).
  3. Usability: how helpful they perceive the strategy to be for them (0 = not at all, to 5 = very).
  The total score for each of the 3 domains are divided by the number of strategies, to reach a mean score for each of the three domains. Results will be examined at a qualitative level to guide further refinement of the intervention.
General Anxiety Disorder -7 | Weekly from baseline to 14 weeks.
  This 7-item version of the GAD questionnaire is a short measure of symptoms of anxiety. Participants are asked how often they have been bothered by a set of anxiety symptoms the last 2 weeks ranging from 0=not at all, to 7=daily. The measure will serve as a control variable in mediation analyses.
Time with high blood glucose | From baseline until 26 weeks.
  Percentage of time the past 2 weeks when blood glucose levels have reached above 13.9 mmol/l. This data will be gathered via the Glooko online glucose system.
Time with high blood glucose (repeated measures) | Every second week from baseline until 14 weeks.
  Percentage of time the past 2 weeks when blood glucose levels have reached above 13.9 mmol/l. This data will be gathered via the Glooko online glucose system.
Blood glucose variation (repeated measures) | Every second week from baseline until 14 weeks.
  Standard deviation of blood glucose levels during the past 2 weeks. This data will gathered via the Glooko online glucose system.
Mean glucose level (repeated measures) | Every second week from baseline until 14 weeks.
  The mean glucose level during the past 2 weeks. This data will be gathered via the Glooko online glucose system.
Time in Target (TiT) (repeated measures) | Every second week from baseline until 14 weeks.
  TiT is the percentage of time that blood glucose levels have been within the target interval 4-8 mmol/l during the last 2 weeks. This data will be gathered via the Glooko online glucose system.
Time with low blood glucose (repeated measures) | Every second week from baseline until 14 weeks.
  Percentage of time during the past two weeks when blood glucose values have reached below 3 mmol/l. This data will be gathered via the Glooko online glucose system.

CONTACTS AND LOCATIONS:
Overall Officials: Brjánn Ljótsson, Professor, Principal Investigator — Karolinska Institute, Department of Clinical Neuroscience, Division of Psychology
Locations (1):
- Karolinska University Hospital, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: No
European GDPR regulation prevents sharing of IDP

DOCUMENTS (1):
  • Statistical Analysis Plan (2025-01-10): https://cdn.clinicaltrials.gov/large-docs/40/NCT06599840/SAP_000.pdf